CLINICAL TRIAL: NCT07136662
Title: How to Improve the Diagnosis of Anderson-Fabry Disease - the Power of Knowledge.
Brief Title: Anderson Fabry Disease - the Power of Information.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Graziani Francesca, DR, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3924
Record Dates: First submitted 2023-02-24; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- learning cardiologist (Other): there will be no arm as the intervention of the study is educational. The promoting centre will enroll other centres with no expertise in rare diseases and will provide targeted information on Fabry cardiomyopathy via webinar.
  The number of patients diagnosed with Fabry disease before and after the study will be the main endpoint
  Interventions: Other: educational

INTERVENTIONS:
Other: educational — see arm description

SUMMARY:
The goal of this before-after control-impact study is to determine whether providing targeted information on Fabry disease (FD) to cardiologists and tutoring them in the evaluation of patients with unexplained left ventricle hypertrophy may improve FD screening and increase FD diagnosis.

Participants (italian cardiologists from centres not experienced in cardiomyoopathies) will be given targeted information on FD viaa training course organized in two parts: a "Theoretical phase" based on on-line interactive lessons on FD and a "Tutored phase" in which the cardiologists from spoke Centers will be actively supported in the diagnostic process.

DETAILED DESCRIPTION:
Background: In Fabry disease (FD), cardiac involvement is frequent and has strong prognostic implications. The main expression of Fabry cardiomyopathy (FC) is left ventricular hypertrophy, mimicking sarcomeric hypertrophic cardiomyopathy. Misdiagnosis is frequent and is mainly related to the lack of knowledge of rare diseases such as FD. Diagnostic delay has a significant prognostic impact in FD since Enzyme Replacement Therapy effects critically depend on the stage of the disease.

Objectives: To determine whether providing targeted information on FD to cardiologists and tutoring them in the evaluation of patients with unexplained LVH may improve FD screening, contributing to reduce both diagnostic and therapeutic delay.

Design of the study: This will be an investigator-initiated research, designed as before-after control-impact study aiming at comparing the rate of FD diagnosis before and after providing targeted information on FD to a group of Italian cardiologist from 54 spoke Centres without outpatient clinics dedicated to cardiomyopathies and with no expertise in rare diseases. The coordinator Centre (Fondazione Policlinico Universitario "A. Gemelli", Rome, Italy) will provide a training course organized in two parts: a "Theoretical phase" based on on-line interactive lessons on FD and a "Tutored phase" in which the cardiologists from spoke Centers will be actively supported in the "diagnostic process" providing them interpretative assistance of ECG and echocardiograms.

Primary outcome: to increase the rate of Fabry disease diagnosis. Statistical analyses: Descriptive statistics will be used to quantitatively describe and summarize the basic characteristics of the study data. A comparison will be made between the rate of screening test and confirmed diagnosis pre and post the provided targeted information on FD and the tutored phase.

ELIGIBILITY:
Inclusion Criteria:

Patients with hypertrophic cardiomyopathy and features suggestive of possible Anderson-Fabry disease, defined as one of the following:

* Patients with left ventricular hypertrophy (LVH) of unknown aetiology (diagnosed in/after the 3rd decade of life) defined by a wall thickness≥13 mm measured on echocardiography or cardiac magnetic resonance, in absence of male-to-male transmission and co-existent pathologies that could explain the increased LV wall thickness (i.e. hypertension, aortic stenosis);
* Patients with LVH (diagnosed in/after the 3rd decade of life) and ECG findings frequently encountered in Fabry cardiomyopathy (short PR interval with high QRS voltage, remarkable repolarization abnormalities..);
* Patients with unexplained LVH (diagnosed in/after the 3rd decade of life) and previous history of stroke, renal failure or clinical characteristics compatible with FD multiorgan involvement.

Exclusion Criteria:

NA

Max Age: 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
FD diagnosis | 6 months
  Absolute and relative number of diagnosis of Anderson Fabry disease

CONTACTS AND LOCATIONS:
Overall Officials: francesca graziani, Principal Investigator — FPG
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided